CLINICAL TRIAL: NCT05861089
Title: Rest PETCO2 As a Predictor of Post-operative Complications in Patient Undergoing Major Vascular Surgery
Brief Title: Rest PETCO2 As a Predictor of Post-operative Complications
Status: Recruiting | Type: Observational
Sponsor: St. Anne's University Hospital Brno, Czech Republic (Other)
Responsible Party: Principal Investigator, Ivan Cundrle, Clinical Professor, St. Anne's University Hospital Brno, Czech Republic
Other Study IDs: 17V/2023
Record Dates: First submitted 2023-05-06; First posted 2023-05-16 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Post-Op Complication
Keywords: vascular surgery; cardiopulmonary exercise testing; end-tidal CO2
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- vascular surgery candidates: End-tidal CO2 will be measured day before surgery. Post-operative cardiovascular and pulmonary complications will be monitored fron the hospital stay, or first 30 days.
  Interventions: Diagnostic Test: end-tidal CO2 measurement

INTERVENTIONS:
Diagnostic Test: end-tidal CO2 measurement — Measurements will take place day before surgery, under resting conditions (while sitting in a quiet room with no disruptions) using the Capnography monitor from Nonin Medical (breath by breath data will be recorded and analyzed). Patients will be allowed to get used to the nasal cannula for the first two minutes. Mean end-tidal CO2 value will then be calculated from the following two minutes of spontaneous breathing.

SUMMARY:
Cardiopulmonary exercise testing (CPET) is considered to be a golden standard in preoperative risk assessment and stratification of high risk patients scheduled for major surgery. However, not all of the patients requiring surgery are willing or able to complete this type of testing.

Vascular surgery patients are predominantly elderly people, with significant comorbidity and high degree of frailty and often can not undergo CPET. In recent years, new parameters with similar prognostic value as standard CPET parameters were studied. Specifically, the partial pressure of end-tidal carbon dioxide (PETCO2) at rest has been shown to have the same prognostic value as ventilatory efficiency.

We hypothesized low PETCO2 at rest will be associated with the development of pulmonary and cardiovascular post-operative complications in patients after major vascular surgery. Accordingly, our aim is to compare PETCO2 measured at rest before surgery in patients who develop post-operative complications and in those who do not.

DETAILED DESCRIPTION:
Cardiopulmonary exercise testing (CPET) is considered to be a golden standard in preoperative risk assessment and stratification of high risk patients scheduled for major surgery. However, not all of the patients requiring surgery are willing or able to complete this type of testing. Moreover, inability to perform CPET has been linked with inferior outcomes following surgery.

Vascular surgery patients are predominantly elderly people, with significant comorbidity and high degree of frailty. Therefore, CPET as a mean of risk stratification would be of an especial interest in this group of patients. However, vascular surgery patients often present with peripheral arterial disease, which may contribute to early leg ischemia during exercise and therefore invalid cardiorespiratory reserve function measurement.

In recent years, new parameters with similar prognostic value as standard CPET parameters were studied. Specifically, the partial pressure of end-tidal carbon dioxide (PETCO2) at rest has been shown to have the same prognostic value as ventilatory efficiency in the prediction of post-operative complications in lung resection surgery patients. Whether the same parameter can be used to predict postoperative complications in a different sub-set of surgical patients (i.e. vascular surgery patients) is yet to be determined.

We hypothesized low PETCO2 at rest will be associated with the development of pulmonary and cardiovascular post-operative complications in patients after major vascular surgery. Accordingly, our aim is to compare PETCO2 measured at rest before surgery in patients who develop post-operative complications and in those who do not.

ELIGIBILITY:
Inclusion Criteria:

* indication for major vascular surgery (aortobifemoral bypass surgery)

Exclusion Criteria:

* tracheostomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients scheduled for vascular surgery will be recruited. This subset of patients was chosen as it usually presents with a number of serious comorbidities and short claudication interval which makes them indicated to, but unable to complete the standard CPET
Sampling Method: Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
pulmonary complications | first 30-post operative days
  post-operative complications
post-operative complications | first 30-post operative days
  cardiovascular complications

SECONDARY OUTCOMES:
hospital length of stay | up to 30 days
  hospital length of stay
intensive care unit length of stay | up to 30 days
  intensive care unit length of stay
mortality | from the first 30-post operative days
  mortality

CONTACTS AND LOCATIONS:
Overall Officials: Ivan Cundrle, MD, PhD, Principal Investigator — St. Anne's University Hospital
Locations (1):
- St. Anne's University Hospital in Brno, Brno, Czech Republic, Czechia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Albouaini K, Egred M, Alahmar A, Wright DJ. Cardiopulmonary exercise testing and its application. Postgrad Med J. 2007 Nov;83(985):675-82. doi: 10.1136/hrt.2007.121558. PMID 17989266
- [Background] Keteyian SJ, Isaac D, Thadani U, Roy BA, Bensimhon DR, McKelvie R, Russell SD, Hellkamp AS, Kraus WE; HF-ACTION Investigators. Safety of symptom-limited cardiopulmonary exercise testing in patients with chronic heart failure due to severe left ventricular systolic dysfunction. Am Heart J. 2009 Oct;158(4 Suppl):S72-7. doi: 10.1016/j.ahj.2009.07.014. PMID 19782792
- [Background] Lai CW, Minto G, Challand CP, Hosie KB, Sneyd JR, Creanor S, Struthers RA. Patients' inability to perform a preoperative cardiopulmonary exercise test or demonstrate an anaerobic threshold is associated with inferior outcomes after major colorectal surgery. Br J Anaesth. 2013 Oct;111(4):607-11. doi: 10.1093/bja/aet193. Epub 2013 Jun 5. PMID 23744818
- [Background] Ambler GK, Kotta PA, Zielinski L, Kalyanasundaram A, Brooks DE, Ali A, Chowdhury MM, Coughlin PA. The Effect of Frailty on Long Term Outcomes in Vascular Surgical Patients. Eur J Vasc Endovasc Surg. 2020 Aug;60(2):264-272. doi: 10.1016/j.ejvs.2020.04.009. Epub 2020 May 14. PMID 32417030
- [Background] Barkat M, Key A, Ali T, Walker P, Duffy N, Snellgrove J, Torella F. Effect of treatment of peripheral arterial disease on the onset of anaerobic exercise during cardiopulmonary exercise testing. Physiol Rep. 2021 Apr;9(7):e14815. doi: 10.14814/phy2.14815. PMID 33818006
- [Background] Brat K, Homolka P, Merta Z, Chobola M, Heroutova M, Bratova M, Mitas L, Chovanec Z, Horvath T, Benej M, Ivicic J, Svoboda M, Sramek V, Olson LJ, Cundrle I Jr. Prediction of Postoperative Complications: Ventilatory Efficiency and Rest End-tidal Carbon Dioxide. Ann Thorac Surg. 2023 May;115(5):1305-1311. doi: 10.1016/j.athoracsur.2021.11.073. Epub 2022 Jan 21. PMID 35074321
- [Background] Brat K, Tothova Z, Merta Z, Taskova A, Homolka P, Vasakova M, Skrickova J, Sramek V, Olson LJ, Cundrle I Jr. Resting End-Tidal Carbon Dioxide Predicts Respiratory Complications in Patients Undergoing Thoracic Surgical Procedures. Ann Thorac Surg. 2016 Nov;102(5):1725-1730. doi: 10.1016/j.athoracsur.2016.05.070. Epub 2016 Aug 3. PMID 27496629
- [Background] Patel SK, Surowiec SM. Intermittent Claudication. 2023 Jul 10. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK430778/ PMID 28613529